CLINICAL TRIAL: NCT06145178
Title: A Phase I First in Human Study to Assess Safety and Immunogenicity of the Human Cytomegalovirus Vaccine Candidate SPYVLP01 With and Without Adjuvants in Healthy Adult Volunteers
Brief Title: A Study of Human Cytomegalovirus (HCMV) Vaccine SPYVLP01 With and Without Adjuvants
Acronym: SPYVAC01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SpyBiotech Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: SPYVAC01
Record Dates: First submitted 2023-11-14; First posted 2023-11-24 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1 (Experimental): Low dose SPYVLP01 alone
  Interventions: Biological: SPYVAC01
- Group 2 (Experimental): High dose SPYVLP01 alone
  Interventions: Biological: SPYVAC01
- Group 3 (Experimental): Low dose + Alhydrogel
  Interventions: Biological: SPYVAC01
- Group 4 (Experimental): High dose + Alhydrogel
  Interventions: Biological: SPYVAC01
- Group 5 (Experimental): Low dose + Matrix-M
  Interventions: Biological: SPYVAC01
- Group 6 (Experimental): High dose + Matrix-M
  Interventions: Biological: SPYVAC01

INTERVENTIONS:
Biological: SPYVAC01 — Novel vaccine SPYVLP01

SUMMARY:
The main purpose of the study is to evaluate the safety and immunogenicity of SPYVLP01 in two different doses with and without adjuvants in healthy adults aged 18-50 years old.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adult volunteers aged 18 to 50 years with a body mass index (BMI) of 19 to 32 kg/m2
* Written informed consent before initiation of any study-specific procedures
* Willing and able to understand and comply with study requirements
* Women of childbearing potential must have a negative pregnancy test at screening and prior dose 1 of vaccine.
* Women of childbearing potential must agree to practice a highly effective form of contraception continuously until 90 days after receiving the last immunization.
* Women of childbearing potential must agree not to donate eggs from screening visit and continuously until 90 days after receiving the last immunization
* Men must agree to practice a highly effective form of contraception with their female partner of childbearing potential from screening visit and continuously until 90 days after receiving the last immunization
* Men must be willing to refrain from sperm donation, from screening visit and continuously until 90 days after receiving the last immunization
* All participants must agree not to be vaccinated with any vaccine other than the study vaccine during the study, starting after screening visit and continuously until 28 days after receiving the last immunization

Exclusion Criteria

* Any acute illness, with or without fever within 72 hours prior to the first immunization
* Pregnancy, lactation, or intention to become pregnant during the study
* Have a known allergy, hypersensitivity, or intolerance to the planned Investigational Medicinal Product (IMP), adjuvants, and including any excipients of the IMP
* Have any medical condition or any major surgery within the past 5 years which could compromise their well-being if they participate in the study, or that could prevent, limit, or confound the protocol-specified assessments
* Have any surgery planned during the study, starting after screening and continuously until at least 90 days after receiving the last immunization
* Any confirmed or suspected immunosuppressive or immunodeficient state and chronic immunosuppressant medication within the past 6 months
* Received any live or inactivated vaccination within 6 months prior to screening or other vaccinations within the 28 days prior to screening
* Have a history of hypersensitivity or serious reactions to previous vaccinations or a history of Guillain-Barré Syndrome within 6 weeks following a previous vaccination
* Had administration of any immunoglobulins and/or any blood products within the 3 months prior to screening
* Had administration of another IMP including vaccines within 90 days or 5 half-lives prior to screening (Visit 1)
* Hepatitis B surface antigen detected in serum at screening
* Seropositive for hepatitis C virus at screening
* Have a history of or suspected immunosuppressive condition, acquired or congenital
* Symptoms of COVID-19 within 30 days prior to screening
* Alcohol or substance abuse that might interfere with the study conduct or completion
* Consume more than 25 units of alcohol per week
* Concurrent involvement in another clinical study or planned involvement during the study period
* Prior receipt of an investigational vaccine
* History of narcolepsy
* Any abnormality or permanent body art (e.g., tattoo) that would obstruct the ability to observe local reactions at the injection site
* Have had any blood loss > 450 mL within the 3 months (90 days) prior to screening or plan to donate blood during the study
* Anticipating the need for immunosuppressive treatment within the next 6 months
* Inability to contact the participant's general practitioner to confirm medical history

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
To assess the safety profile of the vaccine with and without adjuvants | ongoing for 12 months
  The specific endpoints for safety will be actively and passively collected data on Adverse Events (AEs). The following parameters will be assessed:
  * Occurrence of solicited local and systemic reactogenicity signs and symptoms for 7 days following each vaccination
  * Occurrence of unsolicited AEs for 28 days following each vaccination
  * Change from baseline for safety laboratory measures for 28 days following each vaccination
  * Occurrence of Serious Adverse Events (SAEs) during the whole study duration
  * Occurrence of Adverse events of special interest (AESIs) during the whole study duration
To assess the reactogenicity profile of the vaccine with and without adjuvants | ongoing for 12 months
  The specific endpoints for reactogenicity will be actively and passively collected data on AEs. The following parameters will be assessed:
  * Occurrence of solicited local and systemic reactogenicity signs and symptoms for 7 days following each vaccination
  * Occurrence of unsolicited AEs for 28 days following each vaccination
  * Change from baseline for safety laboratory measures for 28 days following each vaccination
  * Occurrence of SAEs during the whole study duration
  * Occurrence of AESIs during the whole study Duration

SECONDARY OUTCOMES:
To investigate the pentamer specific binding antibodies and neutralizing antibodies solicited by each arm in seropositive and seronegative healthy male and female adult volunteers | ongoing for 12 months
  Pentamer-specific immunogenicity will be assessed by a variety of immunological assays.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Velocity Bristol, Bristol
  - Medicines Evaluation Unit, Manchester

IPD SHARING:
Plan to Share IPD: No